CLINICAL TRIAL: NCT01744184
Title: A Single-centre, Randomised Controlled Study of Entonox Versus Midazolam Sedation in Gastroscopy.
Brief Title: A Single-centre Study of Entonox Versus Midazolam Sedation in Gastroscopy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Resource issues, Poor recruitment
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENT1
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Patients Requiring Diagnostic Gastroscopy With Sedation
Keywords: gastroscopy; diagnostic; entonox
MeSH Terms: conditions — Disease | interventions — Entonox; Oxygen; Nitrous Oxide; Midazolam; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam (Active Comparator): midazolam sedation combined with pharyngeal anaesthesia
  Participants randomized to receive midazolam will have an intravenous cannula sited and, following the administration of xylocaine throat spray as above, will be put into the left lateral position. They will then be given up to 5mg midazolam as appropriate to achieve conscious sedation as for standard protocol in endoscopy.
  Interventions: Drug: Midazolam
- Entonox (Experimental): Entonox combined with pharyngeal anaesthesia.
  Pharyngeal anaesthesia, given as 8-16 sprays of xylocaine to the pharynx; 3 minutes will be given to allow the pharynx to become anaesthetized.
  Participants randomized to receive Entonox will be given the 50:50 nitrous oxide:oxygen mix via a mouthpiece with a demand valve system, once in position for the procedure. Inhalations will be given for 3-5 minutes (or until the participant feels adequately sedated) measured using a stopwatch. Oxygen will be given at 2 litres per minute via nasal cannulae during the procedure, (standard care for sedated procedures). The endoscopist will then proceed to intubate the cricopharynx and perform the procedure in the standard manner.
  Interventions: Drug: Entonox

INTERVENTIONS:
Drug: Entonox — Entonox arm
  Other Names: Oxygen 50.0% +/- 2.0%; Nitrous oxide 50.0% +/- 2.0%
  Arms: Entonox
Drug: Midazolam — up to 5mg midazolam as appropriate
  Other Names: Midazolam 1mg/ml Solution for Injection
  Arms: Midazolam

SUMMARY:
This study aims to determine whether Entonox (gas and air) is at least as good as intravenous midazolam in providing analgesia and sedation during gastroscopy. Entonox is used as an adjunct in lower gastrointestinal procedures but is not routinely used in gastroscopy, and there is only one similar published study to date, which was performed in children. The main advantage of Entonox over midazolam is the quick recovery time following withdrawal of the agent, which enables patients to return to independent normal life. The investigators would like to be able to offer Entonox to patients as an option for sedation during gastroscopy, this study is being conducted to determine if it is a safe and feasible option.

ELIGIBILITY:
Inclusion Criteria:

* Male/female aged 18 years or over
* Confirmed clinical requirement to undergo diagnostic gastroscopy
* Suitable for sedation
* Able to provide informed consent

Exclusion Criteria:

* History of chronic respiratory or significant cardiac disease
* Requirement for longer procedure eg Barrett's surveillance
* Previous known adverse reaction to Entonox
* Entonox use in previous 4 days
* Known current vitamin B12 or folate deficiency
* Unable to provide consent
* Any known contraindication to Entonox:
* Gas trapped in a part of the body where its expansion may be dangerous, such as air lodged in an artery or artificial traumatic or spontaneous pneumothorax (collapsed lung).
* Decompression sickness (the bends) or following a recent dive
* Air encephalography
* Severe bullous emphysema
* Myringoplasty
* Gross abdominal distension
* Recent severe injuries to the face and jaw
* Current or recent head injuries
* If the patient has recently had any eye surgery where injections of gas have been used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon McLaughlin, MD, Principal Investigator — The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust
Locations (1):
- The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth, Dorset, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Midazolam: midazolam sedation combined with pharyngeal anaesthesia
  Participants randomized to receive midazolam will have an intravenous cannula sited and, following the administration of xylocaine throat spray as above, will be put into the left lateral position. They will then be given up to 5mg midazolam as appropriate to achieve conscious sedation as for standard protocol in endoscopy.
  Midazolam: up to 5mg midazolam as appropriate
- Entonox: Entonox combined with pharyngeal anaesthesia.
  Pharyngeal anaesthesia, given as 8-16 sprays of xylocaine to the pharynx; 3 minutes will be given to allow the pharynx to become anaesthetized.
  Participants randomized to receive Entonox will be given the 50:50 nitrous oxide:oxygen mix via a mouthpiece with a demand valve system, once in position for the procedure. Inhalations will be given for 3-5 minutes (or until the participant feels adequately sedated) measured using a stopwatch. Oxygen will be given at 2 litres per minute via nasal cannulae during the procedure, (standard care for sedated procedures). The endoscopist will then proceed to intubate the cricopharynx and perform the procedure in the standard manner.
  Entonox: Entonox arm
Period: Overall Study
Arm/Group | Midazolam | Entonox
Started | 32 | 30
Completed | 31 | 29
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Entonox | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants] — Age was not collected. All participants were 18 or over to be eligible for the study. Population: Age was not collected. All participants were 18 or over to be eligible for the study.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Mild or no Discomfort During Gastroscopy
Description: Percentage of patients with a score of 4 or 5 on the 5-point modified global rating scale comfort score, as measured by the patient, will be compared between the midazolam and entonox groups, per protocol. The comfort score ranges from 1-5 with 1 meaning patient was in extreme discomfort frequently during procedure and 5 being no discomfort, resting comfortably throughout. The score is completed by the patient while they are in the recovery area post procedure and prior to discharge from the unit.
Time Frame: During gastroscopy procedure
Measure: Number; unit: percentage of participants
Arm/Group | Midazolam | Entonox
Number analyzed (Participants) | 32 | 30
percentage of participants | 87.5 | 63.3

2. Secondary Outcome: Number of Participants With Completed Procedures in Both Arms of the Study.
Description: The percentage of participants with completed procedures in both arms of the study confirmed by data collection.
Time Frame: Day of procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Midazolam | Entonox
Number analyzed (Participants) | 32 | 30
Percentage of participants | 100 | 96.7

3. Secondary Outcome: Comparison of Procedure Time
Description: Comparison of procedure time, defined as start time to end time in the per protocol population, between the two groups.
Time Frame: Defined as start time to end time of gastroscopy.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Midazolam | Entonox
Number analyzed (Participants) | 32 | 30
Minutes | 4 [3 to 14] | 5 [2 to 19]

4. Secondary Outcome: Comparison of Procedure Start Time to Discharge.
Description: Comparison of gastroscopy procedure start time to discharge from endoscopy department post-procedure care time in the per protocol population between the two groups.
Time Frame: Procedure to discharge
Measure: Median (Full Range); unit: Minutes
Arm/Group | Midazolam | Entonox
Number analyzed (Participants) | 32 | 30
Minutes | 86 [20 to 217] | 46 [16 to 143]

5. Secondary Outcome: Number of Patients With Adverse Events.
Description: Number of patients reporting adverse events.
Time Frame: Consent to 72 hours post discharge from the endoscopy unit which is the same day as the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Entonox
Number analyzed (Participants) | 32 | 30
Participants | 1 | 2

6. Secondary Outcome: Comparison of Visual Analogue Scale Scores.
Description: Comparison of VAS (Visual Analogue Scale) scores between the two groups (per protocol). The scale ranges between 0 and 100 where 0 is the worst imaginable experience and 100 being very comfortable. The visual measure is a 100mm line and the score is measured by the participant marking on the line how they felt the procedure was. The research team then measure the line and confirm the score to the nearest mm to get a score of 0-100.
Time Frame: Completed after procedure completion during the post-procedure care and prior to discharge from the endoscopy unit.
Population: 1 participant in the Midazolam cohort did not complete the Visual Analogue Scale post procedure prior to discharge.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Midazolam | Entonox
Number analyzed (Participants) | 31 | 30
score on a scale | 90 [20 to 100] | 80 [20 to 100]

7. Secondary Outcome: 5-point Modified Global Rating Scale Comfort Nurse Score
Description: Percentage of patients with a score of 4 or 5 on the 5-point comfort scale, as measured by the endoscopy nurse, will be compared between the midazolam and Entonox groups, per protocol. The comfort score ranges from 1-5 with 1 meaning patient was in extreme discomfort frequently during procedure and 5 being no discomfort, resting comfortably throughout. This score is completed by the endoscopy nurse immediately following the patients procedure.
Time Frame: Completed after procedure completion during the post-procedure care and prior to discharge from the endoscopy unit.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam | Entonox
Number analyzed (Participants) | 32 | 30
Participants | 31 | 28

ADVERSE EVENTS:
Time Frame: From participant consent until 72 hours post procedure. Adverse events were monitored while the patient was on site following consent until they were discharged from the endoscopy unit. A follow up phone call was completed 72 hours after the participant was discharged and the participants were asked to recall any adverse events that have occurred since their discharge.
Arm/Group | Midazolam | Entonox
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 1/32 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=32) | Entonox (N=30)
Allergic Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Allergic reaction to cannula plaster
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)
Shivering (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT01744184/Prot_SAP_000.pdf